CLINICAL TRIAL: NCT00711503
Title: A Randomised Clinical Trial of the Effect of Interleukin-1 Receptor Antagonism on the Insulin Production in Patients With New Onset Type 1 Diabetes
Brief Title: Anti-Interleukin-1 in Diabetes Action
Acronym: AIDA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Oeresund Diabetes Academy (Unknown)
Responsible Party: Principal Investigator, Lise Tarnow, professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-007146-34; EudraCT 2007-007146-34; Danish EthicalH-D-2008-060; Danish Datatilsyn2007-41-1652; JDRF file no. 17-2007-1804
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Type 1 Diabetes
Keywords: endogenous insulin production; C-peptide level; insulin requirement
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): The patients are instructed to administer placebo by subcutaneous injection
  Interventions: Drug: saline
- 1 (Experimental): The patients are instructed to administer anti-IL-1 therapy in the form of recombinant human non-glycosylated interleukin-1 receptor antagonist (IL-1Ra, anakinra, Kineret®, Amgen, CA, USA) [13] at a dose of 100 mg once daily by subcutaneous injection
  Interventions: Drug: anakinra

INTERVENTIONS:
Drug: anakinra — The patients are instructed to administer anti-IL-1 therapy in the form of recombinant human non-glycosylated interleukin-1 receptor antagonist (IL-1Ra, anakinra, Kineret®, Amgen, CA, USA) [13] at a dose of 100 mg once daily by subcutaneous injection
  Other Names: Kineret
  Arms: 1
Drug: saline — The patients are instructed to administer placebo (saline) once daily by subcutaneous injection
  Arms: 2

SUMMARY:
A draw trial of the effect of Interleukin-1 Receptor Antagonist (anakinra, Kineret®) on the insulin production in patients with new onset Type 1 diabetes.

Kineret® is already being used in the treatment of patients suffering from rheumatoid arthritis and preclinical studies are now suggesting that it may also be useful for patients with Type 1 diabetes. The active substance in Kineret is interleukin-1 receptor antagonist, a blocker of an immune-signal molecule named interleukin-1.

The trial is a blinded randomised trial, in which the patient is allocated to receive the active drug (Kineret®) or placebo (saline). The hypothesis is that anti-IL-1 treatment as add-on therapy to conventional insulin therapy will preserve or enhance beta-cell function.

DETAILED DESCRIPTION:
Objectives:

The aim of the Anti-Interleukin-1 in Diabetes Action trial (AIDA) study is to test the feasibility, safety/tolerability and potential efficacy of anti-IL-1 therapy in maintaining or enhancing beta-cell function in people with new onset Type 1 diabetes.

Trial Design:

A randomized, placebo controlled, double masked, parallel group, multicentre trial of IL-1 antagonism in subjects with newly-diagnosed Type 1 diabetes. Patients are instructed to inject 100 mg human recombinant interleukin-1 receptor antagonist (anakinra, Kineret®, Amgen, CA) or placebo s.c. once daily for 2 years. Endpoints will be evaluated every three months, with an interim analysis after 6 months.

Trial population:

The design will be a two-stage phase 2a study to address feasibility, safety/tolerability and potential efficacy. In the first phase 80 patients between 18 and 35 years of age with new on-set Type 1 diabetes will be randomized to anakinra or placebo, and endpoints will be analyzed as an interim analysis after 6 months by an independent data and safety monitoring board (DSMB). A futility analysis will be performed at this time point to prevent continuation of the trial if it shows no likelihood of demonstrating efficacy. In the event the trial does show promise of efficacy considering the power of the first phase based on a conditional analysis the DSMB can recommend prolongation of the study with recruitment to ensure adequate power, and that additional funding is provided.

Methods and interventions:

The patients are instructed to administer anti-IL-1 therapy in the form of recombinant human non-glycosylated interleukin-1 receptor antagonist (anakinra) at a dose of 100 mg once daily or placebo by subcutaneous injection at the same time-point in the morning. Primary and secondary endpoints and safety parameters are investigated after 1 month and then every 3 months.

Safety:

Anakinra is FDA approved for the indication rheumatoid arthritis and has an acceptable risk / benefit profile in this indication, with more than 100.000 patients treated. Most common ad-verse events include mild and transient local injection reactions in 20-50% of subjects treated with Anakinra. Consistent with its mechanism of action, anakinra reduces WBC/ANC in 2.4% of patients and this may increase the risk of infection. Accordingly, treatment with anakinra will not be initiated in patients with active infections. Safety will be monitored by physical exams and blood and urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed according to WHO 1999 criteria
* Positive GAD auto-antibodies
* Age 18-35 yrs at onset of diabetes
* Time from first symptoms of diabetes < 12 weeks
* Peak C-peptide more than or equal to 200 pM after a standardized mixed meal test (Boost) at a test carried out when the subject is metabolically stable, i.e. after resolution of any polyuria, polydypsia or ketoacidosis.

Exclusion Criteria:

* Severe liver or renal disease (creatinine > 100 μmol/L, ASAT/ALAT > 2* ULN, alkaline phosphatase > 2 * ULN)
* History of heart disease, signs of cardiac failure or abnormal ECG
* Present or previous malignancy
* Pregnancy or failure of fertile female to comply with contraceptional planning, or breast-feeding. (Safe contraceptive methods include birth control pills, IUD, and gestagen implants) . Plans of pregnancy within 2 years.
* Participation in other clinical intervention studies
* Anti-inflammatory therapy (except aspirin £ 100 mg/d)
* Active infections (CRP>30), history of recurrent infection or predisposition to infections
* Neutropenia: ANC < 1.5*109/L, or anaemia: Haemoglobin < 8.0 g/dL
* Immune-suppressive treatment or immune-deficiency
* Presence at diagnosis of late diabetic complications
* Concurrent vaccination with live vaccine. Known need for live vaccinations within 2 years.
* Use of Etanercept within 6 months before screening or during the double-blinded study period
* Hypersensitivity to E. coli-derived proteins, anakinra or any components of the product.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Δ 2-h AUC C-peptide response | 1 month, 3 months, 6 months, 9 months

SECONDARY OUTCOMES:
Incremental and/or peak C-peptide response, Time to peak C-peptide, insulin requirement per kg body weight per day,frequency of insulin free state with maintenance of HbA1c <7.5%, HbA1c, Means of fasting glucose values, circulating IL-6 and CRP | 1 month, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Mandrup-Poulsen, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen; Marc Donath, Study Director — Universtity of Zürich; Flemming Pociot, DMSc, Study Director — Steno Diabetes Center Copenhagen; Charles Dinarello, Study Director — University of Colorado Health Science Center; Edwin Gale, Professor, Study Chair — Bristol University, UK
Locations (17):
- Denmark (5):
  - Aalborg Hospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Universitetshospital, Copenhagen
  - Steno Diabetes Center, Gentofte Municipality
  - Nordsjællands Hospital, Hillerød, Hillerød
- Germany (4):
  - Ulm University, Dept. of Internal Medicine, Ulm, Donau
  - Leibniz Center for Diabetes research, Heinrich-Heine University, Düsseldorf
  - University of Frankfurt am Main, Frankfurt am Main
  - Institut für Diabetesforschung, Munich University of Technology, Munich
- University Campus Bio-Medico, Rome, Italy
- Leiden University Medical Center, Leiden, Netherlands
- Medical University of Bialystok, Bialystok, Poland
- Spain (4):
  - Hospital de Cruces, Diabetes Research Group, Barakaldo, Bizkaia
  - Hospital Unversitario Insular de Gran Canaria, Las Palmas, Gran Canaria
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Arnua de Vilanova, Lleida
- University Hospital Zürich, Zurich, Switzerland

REFERENCES:
- [Background] Pickersgill LM, Mandrup-Poulsen TR. The anti-interleukin-1 in type 1 diabetes action trial--background and rationale. Diabetes Metab Res Rev. 2009 May;25(4):321-4. doi: 10.1002/dmrr.960. PMID 19405081
- [Derived] Moran A, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Greenbaum CJ, Herold KC, Marks JB, Raskin P, Sanda S, Schatz D, Wherrett DK, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Canakinumab Study Group; Pickersgill L, de Koning E, Ziegler AG, Boehm B, Badenhoop K, Schloot N, Bak JF, Pozzilli P, Mauricio D, Donath MY, Castano L, Wagner A, Lervang HH, Perrild H, Mandrup-Poulsen T; AIDA Study Group. Interleukin-1 antagonism in type 1 diabetes of recent onset: two multicentre, randomised, double-blind, placebo-controlled trials. Lancet. 2013 Jun 1;381(9881):1905-15. doi: 10.1016/S0140-6736(13)60023-9. Epub 2013 Apr 5. PMID 23562090